CLINICAL TRIAL: NCT06969027
Title: JS207 (PD-1/VEGF Dual Antibody) Combined With Chemotherapy in First-line Treatment of Advanced Non-small Cell Lung Cancer
Brief Title: JS207Combined With Chemotherapy in First-line Treatment of Advanced NSCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JS207-010-II-NSCLC
Record Dates: First submitted 2025-04-28; First posted 2025-05-13 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Platinum; Paclitaxel

STUDY DESIGN:
Intervention Model Description: Arm 1: JS207 (10 mg/kg or 15 mg/kg, IV, D1) + Pemetrexed (500 mg/m2 IV, D1) + a platinum (carboplatin AUC 5, D1 or cisplatin 75 mg/m2, D1), Q3W, for 4 cycles followed by JS207 (10 mg/kg or 15 mg/kg, IV, D1) + pemetrexed (500 mg/m2 IV, D1), Q3W.
  Arm 2: JS207 (10 mg/kg or 15 mg/kg, IV, D1) + Paclitaxel (175 mg/m2 IV, D1) + a platinum (carboplatin AUC 5, D1 or cisplatin 75 mg/m2, D1), Q3W, for 4 cycles followed by JS207 (10 mg/kg or 15 mg/kg, IV, D1), Q3W.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JS207+ Pemetrexed + a platinum (Experimental): Enrolling 30-42 Non-squamous non-small cell lung cancerparticipants，Patients will receive JS207 (10 mg/kg or 15 mg/kg, IV, D1) + Pemetrexed (500 mg/m2 IV, D1) + a platinum (carboplatin AUC 5, D1 or cisplatin 75 mg/m2, D1), Q3W, for 4 cycles followed by JS207 (10 mg/kg or 15 mg/kg, IV, D1) + pemetrexed (500 mg/m2 IV, D1), Q3W.
  Interventions: Drug: JS207; Drug: Pemetrexed injection; Drug: Platinum
- JS207+ Paclitaxel + a platinum (Experimental): Enrolling 30-42 squamous non-small cell lung cancerparticipants，Patients will receive JS207 (10 mg/kg or 15 mg/kg, IV, D1) + Paclitaxel (175 mg/m2 IV, D1) + a platinum (carboplatin AUC 5, D1 or cisplatin 75 mg/m2, D1), Q3W, for 4 cycles followed by JS207 (10 mg/kg or 15 mg/kg, IV, D1), Q3W.
  Interventions: Drug: JS207; Drug: Platinum; Drug: Paclitaxel

INTERVENTIONS:
Drug: JS207 — JS207 (10 mg/kg or 15 mg/kg, IV, d1)
Drug: Pemetrexed injection — Pemetrexed (500 mg/m2 IV, D1)
  Arms: JS207+ Pemetrexed + a platinum
Drug: Platinum — Platinum (carboplatin AUC 5, D1 or cisplatin 75 mg/m2, D1)
Drug: Paclitaxel — Paclitaxel (175 mg/m2 IV, D1)
  Arms: JS207+ Paclitaxel + a platinum

SUMMARY:
This study targets patients with in first-line treatment of advanced NSCLC， enrolling 60-84 participants. Patients will receive Arm 1: JS207 (10 mg/kg or 15 mg/kg, IV, D1) + Pemetrexed (500 mg/m2 IV, D1) + a platinum (carboplatin AUC 5, D1 or cisplatin 75 mg/m2, D1), Q3W, for 4 cycles followed by JS207 (10 mg/kg or 15 mg/kg, IV, D1) + pemetrexed (500 mg/m2 IV, D1), Q3W, until meeting the treatment withdrawal criteria. Arm 2: JS207 (10 mg/kg or 15 mg/kg, IV, D1) + Paclitaxel (175 mg/m2 IV, D1) + a platinum (carboplatin AUC 5, D1 or cisplatin 75 mg/m2, D1), Q3W, for 4 cycles followed by JS207 (10 mg/kg or 15 mg/kg, IV, D1), Q3W, until meeting the treatment withdrawal criteria.The study aims to assess the safety, tolerability, and preliminary efficacy of JS207 combination therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75 years old (both 18 and 75 years old included) at the time of signing the informed consent form, applicable to both males and females.
2. Locally advanced (stage IIIB/IIIC), metastatic or recurrent non-small cell lung cancer (NSCLC) confirmed by histology or cytology, which is not eligible for radical surgery or radical chemoradiotherapy.
3. History of no systemic antitumor therapy for Metastatic or recurrent NSCLC; for subjects who have received adjuvant/neoadjuvant/consolidation therapy (Chemotherapy, radiotherapy, or other therapy), they can be enrolled if the interval between the last treatment and recurrence is more than 6 months.
4. Tissue samples are required for PD-L1 test. New tissue samples are preferred. If new tissue samples are not available, archived samples can be provided.
5. According to the RECIST v1.1 criteria, the subject has at least 1 measurable lesion.
6. Performance status score of 0-1 according to the Eastern Cooperative Oncology Group (ECOG) scale.
7. Expected survival period ≥ 12 weeks.
8. The function of important organs meets the requirements of the protocol.
9. Female subjects of childbearing potential, and male subjects whose partners are females of childbearing age, need to adopt a highly effective contraceptive measure during the study treatment period and for at least 6 months after the last administration.
10. Voluntarily joining this study, signing the informed consent form, having good compliance, and cooperating with the follow-up.

Exclusion Criteria:

1. Histopathologically or cytopathologically confirmed to have combined neuroendocrine (including small cell lung cancer and large cell neuroendocrine carcinoma) components.
2. Treatment received as listed in the protocol, including immunologically mediated treatment; drugs targeting the anti-VEGF pathway, etc.
3. Having an obvious bleeding tendency or a history of severe coagulation dysfunction.
4. Gastrointestinal perforation, intra-abdominal fistula or intra-abdominal abscess occurred within 6 months before the first administration, or currently having high-risk factors for perforation/fistula formation of the hollow viscus as judged by the investigator.
5. Having a serious, unhealed or ruptured wound, active ulcer or untreated fracture.
6. Having uncontrolled hypertension, or a history of hypertensive crisis or hypertensive encephalopathy.
7. Expected that the toxicity of previous anti-tumor treatment has not recovered to ≤ grade 1 according to the Common Terminology Criteria for Adverse Events (CTCAE).
8. Known allergy to the investigational drug or its excipients, pemetrexed, platinum drugs (carboplatin/cisplatin), or known history of ≥ grade 3 allergy to antibody drugs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-06-19 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Investigator-assessed objective response rate (ORR) | Up to approximately 25 months
  Evaluate the investigator-assessed objective response rate (ORR) of JS207 combined with chemotherapy in the treatment of n first-line treatment of advanced non-small cell lung cancer (NSCLC) patients.The ORR is defined as the proportion of subjects who have a partial response (PR) or a complete response (CR) in the Best Overall Response.

SECONDARY OUTCOMES:
Investigator-assessed objective response rate (DCR) | Up to approximately 25 months
  The DCR is defined as the proportion of subjects whose Best Overall Response (BOR) is Complete Response (CR), Partial Response (PR), or Stable Disease (SD).
Investigator-assessed Progression-Free Survival (PFS) | Up to approximately 25months
  The PFS is defined as the time from the first administration of the drug to the first documented disease progression (PD) according to the RECIST v1.1 criteria or death due to any disease (whichever occurs first).
Investigator-assessed overall survival (OS) | Up to approximately 30 months
  The OS is defined as the time from the first administration of the drug to death due to any cause.
Adverse Event | Up to approximately 25 months
  Collect Serious Adverse Events (SAEs) and Adverse Events (AEs) from the time of signing the Informed Consent Form (ICF) until the safety follow-up visit.Evaluate the safety of the investigational drug.
Abnormal changes in laboratory | Up to approximately 25 months
  Incidence and serverity of abnormal changes in laboratory and other tests with clinical significance

OTHER OUTCOMES:
PK | Up to approximately 25 months
  To characterize the trough concentrations of JS207
Immunogenicity (ADA） | Up to approximately 25 months
  The immunogenicity of JS207, including the incidence rate of anti-drug antibodies (ADA)
Immunogenicity （Nab） | Up to approximately 25 months
  The immunogenicity of JS207, including the incidence rate of neutralizing antibodies (NAb) (if applicable)，the titer of ADA
Expression level of PD-L1 in tumor tissues | Up to approximately 5 months
  Measuring the expression level of PD-L1 Protein in a Neoplasm tissue sample from a subject by an Immunohistochemistry assay

CONTACTS AND LOCATIONS:
Overall Officials: Weihua Wang, Doctor, Study Director — Medical Director
Locations (1):
- Shandong First Medical University Affiliated Neoplasm Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No